CLINICAL TRIAL: NCT03028558
Title: Biology of the Oral Epithelium of E-Cigarette Smokers
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1512016796
Record Dates: First submitted 2017-01-11; First posted 2017-01-23 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Electronic Cigarettes; Healthy Volunteers; E-Cigarettes Smokers; E-Cigarettes
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected may include blood, urine and oral epithelium samples from consenting subjects. Subjects will include both e-cigarette smoking individuals and healthy control subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HEALTHY VOLUNTEER RESEARCH SUBJECTS: Healthy as defined by those not having lung disease and inclusive of: all races, ethnicities, sex, HIV status, smoking status and multiple birth status, etc., within the general population.
  Between the ages of 21-35 years old.
- HEALTHY E-CIGARETTE SMOKING SUBJECTS: Criteria is identical to the healthy never-smoker group except that they must have a history of smoking e-cigarettes >5 days/wk for a minimum of 6 months with no prior traditional tobacco exposure.

SUMMARY:
Electronic cigarettes (EC) are battery powered nicotine delivery devices that aerosolize nicotine and other flavor constituents. Despite the increasing use of EC, little attention has been paid to their possible adverse effects on human health. Theoretically, the risk relates to nicotine per se and/or the propellants or contaminants in the EC aerosol. The hypothesis underlying the proposal is that chronic EC smoking disorders the biology of the oral epithelium, the first cell population exposed to inhaled EC vapors. Using a cross-sectional, cohort-comparison of EC smokers compared to age-, gender- and ethnicity-matched never smokers, the investigators propose to assess the oral epithelium obtained by punch biopsy or brushing from 100 EC smokers and 25 nonsmoker controls. The EC study cohort will be restricted to young adults (age 21-35 yr) with no prior history of tobacco smoking, but who have smoked EC for >6 months.

DETAILED DESCRIPTION:
There is compelling evidence to support this hypothesis: (1) EC vapors contain nicotine, the oral epithelium expresses nicotine receptors, and exposure of epithelia to nicotine activates the nicotine pathway; (2) EC vapors also contain chemical contaminants that can potentially effect oral epithelial biology; and (3) in vitro studies suggest that EC vapors modify epithelial biology and data generated by our laboratory demonstrates that even a brief, acute exposure of healthy nonsmokers to EC vapors induces significant changes in the airway epithelial transcriptome, including the expression of genes in the nicotine and p53 pathways. With the knowledge that disordering of cell biology occurs long before clinical disease,the investigators will evaluate the oral epithelium at the transcriptome (mRNA and miRNA) levels. They will then identify gene(s)/pathways/communities disordered by EC vapors.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY VOLUNTEER RESEARCH SUBJECTS:

Inclusion Criteria:

* Males and females, ages 21 to 35
* Must be capable of providing informed consent
* Self-reported never-smokers of any type, including chewing tobacco, with current smoking status validated by the absence of nicotine metabolites in urine (nicotine <2 ng/ml and cotinine <5 ng/ml)
* No bleeding diathesis
* Normal physical examination
* Good overall health without history of oral or lung disease
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/immunologic studies, general biochemical analyses, and urine analysis
* Not taking any medications relevant to lung disease or having an effect on the airway epithelium
* Normal chest X-ray (PA and lateral)
* Normal electrocardiogram (sinus bradycardia, premature atrial contractions are permissible)
* Females - not pregnant
* Willingness to participate in the study

  * HEALTHY VOLUNTEER E-CIGARETTE SMOKING SUBJECTS:

Inclusion Criteria:

* Males and females, ages 21 to 35
* Must be capable of providing informed consent
* E-cigarette smokers with current smoking status validated by nicotine metabolites in urine (nicotine >20 ng/ml and cotinine >30 ng/ml)
* No bleeding diathesis
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/immunologic studies, general biochemical analyses, and urine analysis
* Good overall health without history of oral disease
* Normal spirometry
* All individuals have chest X-ray (PA and lateral)
* Normal electrocardiogram (sinus bradycardia, premature atrial contractions are permissible)
* Females - not pregnant
* Willingness to participate in the study

Exclusion Criteria:

* HEALTHY VOLUNTEER RESEARCH SUBJECTS:

Exclusion Criteria:

* Unable to meet the inclusion criteria
* Have smoked any form of tobacco
* Current marijuana smokers (within the last three months)
* Current active infection or acute illness of any kind
* Evidence of malignancy, including oral cancer
* Current pregnancy

  * HEALTHY VOLUNTEER E-CIGARETTE SMOKING SUBJECTS:

Exclusion criteria:

* Unable to meet the inclusion criteria
* Have smoked any form of tobacco
* Current marijuana smokers (within the last three months)
* Current active infection or acute illness of any kind
* Evidence of malignancy, including oral cancer
* Current Pregnancy

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators plan recruit the EC smoking (also called "vaping") population, and have experience recruiting from the extensive network of EC shops and vaping "bars" in the New York City metropolitan area, providing ample access to young adult, sole EC smokers. The control groups will be age-, gender- and ethnicity-matched healthy nonsmokers. Based on our experience with this population, the investigators know that the variables of EC smoking history (brand, flavorings, length and extent of EC smoking history) demand that there is sufficient "n" to power the analysis. In this regard, the study population will include n=125, including n=100 EC smokers and a control group of n=25 healthy nonsmokers. Between the ages of 21-35 years old.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
The biology of participants oral epithelial cells | 1-2 months
  Biopsies will be collected from the buccal mucosa of chronic EC smokers and healthy nonsmoker controls, none of whom have a history of smoking any tobacco products

SECONDARY OUTCOMES:
The biology of the genes of the oral epithelium | 1-2 months
  Biopsies will be collected from the buccal mucosa of chronic EC smokers and healthy nonsmoker controls, none of whom have a history of smoking any tobacco products

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Department of Genetic Medicine, Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided